CLINICAL TRIAL: NCT01315808
Title: Rate of Change of HbA1c (dx/dt) May Predict Progression to Type 2 DM: Comparing the Concept of dx/dt With QD Diabetes Prediction Model. D.E.R.M.S Initiative (Doctor Enabled Risk Management System)
Brief Title: Rate of Change of HbA1c (dx/dt) May Predict Progression to Type 2 DM
Status: Terminated | Type: Observational
Why Stopped: Due to lack of funds to continue this study.
Sponsor: Wyckoff Heights Medical Center (Other)
Responsible Party: Rekha Bhandari, Wyckoff Heights Medical Center
Other Study IDs: whmc1
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low risk group: Patients will be stratified based on risk factors significantly contributing to diabetes type 2.
- Intermediate risk group
- High risk group

SUMMARY:
The investigators hypothesize that the HbA1c shows a rising trend in pre-diabetics and normal population with risk factors of developing type 2 DM. There is no known diabetes model for predicting incident diabetes in an individual which takes into account the rate of change of HbA1c (dx/dt). In such cases, the rate of change of HbA1c may give the physicians lead time needed to implement the Diabetes Prevention Program measures.

ELIGIBILITY:
Inclusion Criteria:

* No self-reported history of diabetes or pre-diabetes defined as per ADA criteria
* Age greater than 18 years
* Scheduled to receive HbA1c in participating clinic
* Able and willing to give legally effective consent
* Able and willing to participate in patient questionnaires(attached)

Exclusion Criteria:

* Previously or currently taking medications for lowering glucose (i.e., exenatide, pramlintide, metformin, rosiglitazone, pioglitazone, or future diabetes drugs) based on self-report and/or prescreening. Patients on drugs causing hyperglycemia like Oral Steroids will be excluded.
* Baseline HbA1c level above 5.7
* Severe Anemia (defined as Hb less than 8gm/dL)
* Patients with hemoglobinopathies
* Pregnancy
* Polycystic ovarian disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 1000 non-diabetes people those having at least one diabetes prone risk factor.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Study the rate of change of HbA1c in normal population with known risk factors of diabetes | one year

SECONDARY OUTCOMES:
Diabetes prediction model based on the rate of change in HbA1c | one year
  To develop a mathematical model which will predict the onset of type 2 dm based on the rate of change in HbA1c valued leading to development of pre-diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Bhandari, MD, Principal Investigator — Wyckoff Heights Medical Center, Brooklyn New York; Shitij Arora, MD, Principal Investigator — Wyckoff Heights Medical Center
Locations (1):
- Wyckoff Heights Medical Center, Brooklyn, New York, United States